CLINICAL TRIAL: NCT01226433
Title: Providing Family Planning Services Sustainably Through Dairy Cooperatives in Kenya
Brief Title: Family Planning Through Dairy Cooperatives
Status: Completed | Type: Observational
Sponsor: FHI 360 (Other)
Collaborators: United States Agency for International Development (USAID) (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: 10227
Record Dates: First submitted 2010-10-08; First posted 2010-10-22 (Estimated); Last update posted 2013-03-29 (Estimated); Status verified 2013-03

CONDITIONS: The Study Goal is to Assess the Introduction of Sustainable Family Planning/Reproductive Health Information and Services Through; Land O' Lakes-supported Dairy Cooperatives
Keywords: AE adverse event; AIDS acquired immunodeficiency syndrome; ALT (SGPT) alanine aminotransferase; ART antiretroviral therapy; AST (SGOT) aspartate aminotransferase; DCF data collection forms; DMC Data Monitoring Committee; FDA (U.S.) Food and Drug Administration; GCP Good Clinical Practice guidelines; HB sAg Hepatitis B surface antigen; ICH International Conference of Harmonisation; IND Investigational New Drug Application; IRB Institutional Review Board; IU International units; mg milligram(s); mm3 cubic millimeter(s); PCR polymerase chain reaction; SAE serious adverse event; µg microgram; ULN upper limit of the normal range; WB Western Blot
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

SUMMARY:
This observational study will assess a model for providing family planning through quarterly events organized by dairy cooperatives supported by Land O'Lakes in Kenya.

DETAILED DESCRIPTION:
Access to family planning and other reproductive health services remains difficult in much of rural Kenya. One option for improving rural access to family planning is to use existing community events outside of the health sector as platforms for delivering information and services. This study will assess a model for providing family planning through quarterly events organized by dairy cooperatives supported by Land O'Lakes in Kenya. During these events, known as Field Days, a healthcare provider will have a tent in which Field Day attendees can receive basic family health services free of charge. The services offered will be: family planning counseling and methods, immunizations, antenatal care, screening and treatment for sexually transmitted infections, and HIV counseling and testing. Since the services are no different than those that could be obtained at Ministry of Health or some private facilities, the service provision is not considered to be part of the research.

Women receiving any service from the health care provider will be recruited for an interview that will measure their demand for family planning and attitudes about receiving services during the field day. In addition, the study will track the number of different types of services provided, the total number of Field Day attendees, and the cost of the service model. The study will be carried out at five Field Days in Rift Valley and Central provinces.

Participants will not be tested for STI/HIV as part of this research; however, at their request, they may have received a test from the provider prior to the research interview. At the time of consent, they will have already received the test, so the consent form will not include anything specific to testing. In Kenya, all STI/HIV test results are reported to the national public health authorities. These reports are not used for contacting patients but for planning purposes.

ELIGIBILITY:
Inclusion Criteria:females aged 18-49 receiving health services at a field day event -

Exclusion Criteria:

-

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Females aged 18-49
Sampling Method: Non-Probability Sample
Enrollment: 319 (Actual)
Dates: Start 2010-10; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Health Services Research | 1 year
  Unmet need for family planning among women attending Field Days aged 18-49

SECONDARY OUTCOMES:
Health Services Research | 1 year
  Interest in receiving health services through Field Day model

CONTACTS AND LOCATIONS:
Overall Officials: John Bratt, MPP, MA, Principal Investigator — FHI 360
Locations (1):
- 5 Community Outreach Events, Various, Rift Valley & Central, Kenya